CLINICAL TRIAL: NCT00777309
Title: A Randomized Phase 2 Study of Erlotinib Plus ARQ 197 Versus Erlotinib Plus Placebo in Previously Treated Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Randomized Phase 2 Study of Erlotinib + ARQ 197 Versus Erlotinib + Placebo in Previously Treated Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARQ 197-209
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ARQ 197; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Erlotinib (150 mg) once daily plus ARQ 197 (360 mg) twice daily.
  Interventions: Drug: ARQ 197; Drug: Erlotinib
- 2 (Active Comparator): Erlotinib (150 mg) once daily plus ARQ 197 placebo twice daily
  Interventions: Drug: Erlotinib; Drug: Placebo

INTERVENTIONS:
Drug: ARQ 197 — 360 mg administered twice daily until disease progression, unacceptable toxicity or other discontinuation criterion is met
  Other Names: Tivantinib
  Arms: 1
Drug: Erlotinib — Erlotinib is a white, film coated tablet in strengths of 25, 100 and 150 mg administered once daily until disease progression, unacceptable toxicity or other discontinuation criterion is met.
  Other Names: Tarceva
Drug: Placebo — The placebo is provided as a capsule
  Arms: 2

SUMMARY:
This is a randomized, placebo-controlled, double blind phase 2 study designed to compare treatment with ARQ 197 plus erlotinib to erlotinib plus placebo in patients with non-small cell lung cancer. The study will enroll patients who have had one prior chemotherapy regimen (other than erlotinib) for NSCLC.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double blind phase 2 study designed to compare treatment with ARQ 197 plus erlotinib to erlotinib plus placebo in patients with non-small cell lung cancer. The study will enroll patients who have had one prior chemotherapy regimen (other than erlotinib) for NSCLC. The study will evaluate progression-free survival between the two arms.

A total of 154 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent prior to study-specific screening procedures
2. ≥ 18 years old
3. Histologically or cytologically confirmed inoperable locally advanced or metastatic (stage IIIB/IV) NSCLC
4. ≥ one prior chemotherapy regimen (including adjuvant chemotherapy)(not to have included erlotinib or other EGFR inhibiting agent)
5. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
7. Male or female patients of child-producing potential must agree to use double barrier contraception, oral contraceptives or avoidance of pregnancy measures during the study and for 90 days after the last day of treatment
8. Females of childbearing potential must have a negative serum pregnancy test
9. Good organ function
10. Confirmed availability of archival pathology samples (10 unstained paraffin-embedded slides) or tissue block suitable for subsequent analysis of KRAS, EGFR, and c-Met

Exclusion Criteria:

1. Previous receipt of erlotinib or other EGFR inhibiting therapy
2. Receipt of any anti-tumor treatment for NSCLC within 4 weeks (2 weeks for radiotherapy) prior to the start of designated treatment
3. Documented major surgical procedure within 4 weeks prior to randomization.
4. Symptomatic central nervous system metastases either considered in the opinion of investigator to be clinically unstable or which require steroids, anti-epileptics, or other symptom-relieving medications
5. Pregnant, breast-feeding, or refusing double barrier contraception, oral contraceptives or avoidance of pregnancy measures
6. Significant gastrointestinal disorder that, in opinion of Investigator, could interfere with the absorption of ARQ 197 and/or erlotinib (e.g. Crohn's disease, small or large bowel resection, malabsorbtion syndrome)
7. Unable or unwilling to swallow the complete dose of erlotinib or ARQ 197
8. Any known contraindication to treatment with ARQ 197 or erlotinib
9. Any known hypersensitivity to any of component of ARQ 197 or erlotinib
10. Other malignancy within 5 years of randomization, with the exception of adequately treated intraepithelial carcinoma of the cervix uteri, prostate carcinoma with a PSA value < 0.2 ng/ml or basal or squamous cell carcinoma of the skin
11. Previously diagnosed grade 3 or 4 (CTCAE) bradycardia or other heart arrhythmia
12. Any other significant co-mormid condition that, in opinion of the Investigator, would impair study participation or cooperation
13. Known human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Evaluate progression free survival (PFS) in patients treated with erlotinib plus ARQ 197 versus erlotinib plus placebo

SECONDARY OUTCOMES:
Evaluate overall survival (OS)
Overall response rate (ORR)
Safety of ARQ 197 in combination with erlotinib in patients with NSCLC

CONTACTS AND LOCATIONS:
Locations (36):
- United States (17):
  - Burbank, California
  - Santa Monica, California
  - Torrington, Connecticut
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Batesville, Indiana
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Charlotte, North Carolina
  - Canton, Ohio
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
- Germany (6):
  - Gauting
  - Großhansdorf
  - Hamburg
  - Mainz
  - Mannheim
  - Villingen-Schwenningen
- Latvia (2):
  - Daugavpils
  - Riga
- Poland (6):
  - Bialystock
  - Otwock
  - Poznan
  - Szczecin
  - Torun
  - Wroclaw
- Russia (4):
  - Central Clinical Hospital #1, Moscow
  - Central Clinical Hospital #2, Moscow
  - Saint Petersburg
  - Saint Petersgurg
- Lviv, Ukraine